CLINICAL TRIAL: NCT06691282
Title: A Self-compassion Intervention for LGBTQ+ Individuals: a Feasibility Study
Brief Title: A Self-compassion Intervention for LGBTQ+ Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Polly MA Haixia, Assistant Professor, Hong Kong Metropolitan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HE-RGC2024/NHS14
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-12

CONDITIONS: LGBTQ; Mental Health; Body Image; Self-Compassion
Keywords: LGBT; mental health; self-compassion; body image
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-compassion group (Experimental): Participants in the intervention group will receive 6 weeks self-compassion training.
  Interventions: Other: Mindful self-compassion intervention

INTERVENTIONS:
Other: Mindful self-compassion intervention — Participants will receive six weekly sessions of training by a trainer in mindful self-compassion (MSC). Each session lasting around 90 minutes and will be conducted face-to-face at the Hong Kong Metropolitan University. The content of the intervention will include an introduction of mindfulness and self-compassion, practice of body awareness and loving kindness, skills to deal with challenging experiences, and methods for relating to positive aspects of the self.

SUMMARY:
Gender and sexual minorities often face minority stress, leading to body dissatisfaction and potential psychological issues like anxiety and depression. Self-compassion has been identified as an effective strategy for managing emotions during negative experiences and may serve as a protective factor against minority stress and body image concerns. However, research on self-compassion interventions specifically for LGBTQ+ individuals is limited. This study aims to evaluate the feasibility, acceptability, and preliminary effectiveness of a self-compassion intervention to enhance body image and psychological well-being among LGBTQ+ individuals in Hong Kong.

DETAILED DESCRIPTION:
Gender and sexual minorities often experience minority stress, which could lead to negative thoughts and feelings of their bodies. The substantial body dissatisfaction may contribute to psychological issues such as anxiety and depression. Self-compassion has emerged as an adaptive methods for regulating emotions in response to negative experience and perceived personal failures. Research indicates that self-compassion could act as protective factors of sexual minority stress and body image concerns. However, there is currently a lack of studies investigating the effectiveness of the self-compassion based intervention in improving body image and psychological outcomes among LGBTQ+ individuals.

The proposed study aims to examine the feasibility, acceptability, and preliminary efficacy of a self-compassion intervention for body image and psychological well-being among lesbian, gay, bisexual, transgender and queer (LGBTQ+) individuals in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above;
* Self-identified as LGBTQ+;
* Able to speak, read, and write Cantonese or Putonghua;
* Willing to participate in the study and share their experience of the intervention with the research team;
* Provide written informed consent to participate in the study.

Exclusion Criteria:

* Current psychosis or intellectual disability;
* Current suicidal ideation with intent (score ≥ 4) as measured using the Columbia suicide severity rating scale;
* Participation in similar studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-12-21 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Self-compassion | Through study completion, on average 4 weeks
  Self-compassion, will be measured with the Chinese version of the short version of self-compassion. It has 12 items, and each item is rated on a 5-point Likert scale (1=almost never, 5= almost always). The total score ranged from 12 to 60, with the higher score indicating a higher level of self-compassion.
Internalized stigma | Through study completion, on average 4 weeks
  Internalized stigma will be measured by the Chinese version of the 9-item self-stigma scale, which assesses cognitive, affective, and behavioral components of internalized stigma. The nine items are rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree), with a higher score indicating a higher level of internalized stigma. The scale has shown excellent internal consistency in Chinese sexual minorities, with a Cronbach's alpha ranging from 0.92 to 0.93.

SECONDARY OUTCOMES:
Body image | Through study completion, an average of 4 weeks
  Body image, will be assessed through the Chinese version of the body appreciation scale (BAS-2). It has 10 items, All items are rated on a 5-point Likert scale, ranging from 1 (never) to 5 (always). The total score ranges from 5 to 50, with the higher score representing a higher level of body appreciation.
Anxiety | Through study completion, an average of 4 weeks
  Anxiety, evaluated using the Chinese version of the generalized anxiety disorders (GAD). It has 7 items, each item is rated on a 4-point Liker scale, from 0 (not at all) to 3 (nearly everyday). The total score ranges from 0 to 21, with the higher score representing a higher level of anxiety.
Depression | Through study completion, an average of 4 weeks
  Depression will be measured using the Chinese version of the 9-item patient health questionnaire (PHQ-9). Every item is rated on a 4-point Likert scale, from 0 (not at all) to 3 (nearly everyday). The total score ranges from 0 to 27, with the higher score representing a higher level of depression.
Self-objectification | Through study completion, on average 4 weeks
  Self-objectification will be measured using the body surveillance and body shame subscales of the Chinese version of the Objectified Body Consciousness Scale (OBCS)-body surveillance subscale. The two subscales consist of 14 items. Each item is rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating higher levels of body surveillance and body shame. The Cronbach's alpha for body surveillance was 0.80 for Chinese women and 0.81 for Chinese men, and the Cronbach's alpha for body shame was 0.70 for both Chinese women and men.
self-esteem | Through study completion, on average 4 weeks
  Participants' self-esteem was assessed by the Rosenberg Self-esteem Scale (RES) [25]. The RES is a 10-item scale that measures self-esteem on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The total score is calculated by summing the responses, with higher scores indicating high levels of self-esteem. The Chinese version of RES has demonstrated reliability among PWUD with a Cronbach's α of 0.76.

CONTACTS AND LOCATIONS:
Overall Officials: Haixia Ma, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- School of Nursing and Health Sciences, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
To ensure participant confidentiality, individual data will remain private and will not be shared.